CLINICAL TRIAL: NCT00436878
Title: Intake Promoting Effects of Large Portions in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DK71095; R01DK071095 (NIH)
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Eating
Keywords: Eating Behavior; Children; Portion size; Experimental
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Portion Size (Experimental): Each experiment manipulated food portion size of beverages, entrees, and side dishes
  Interventions: Behavioral: Food portion size

INTERVENTIONS:
Behavioral: Food portion size — Each of four experiments involves a 2 x 2 within-subjects factorial design, in which the first factor is the portion size of a food served to children: foods will be served in a reference amount (i.e. 250 g macaroni and cheese) or doubled in size(i.e. 500 g of macaroni and cheese). In the Experiment 1, the second factor of the 2 x 2 design is meal type: whether the food is consumed at a meal or a snack. In experiment #2, the second factor is food type: fruit vs. vegetable. In experiment #3, the second factor is entree energy density: a regular energy density or a 40% greater energy density. In experiment #4, the second factor is plate size: a 6 inch plate vs. a 10 inch plate.

SUMMARY:
The purpose of this study is to test the effects of large food portions on children's eating. Experiment 1 will test the effect of portion size on children's consumption of sweetened beverages; we hypothesize that serving large beverage portions will increase the amount of energy children consume from this food. Experiment 2 will test the effects of portion size on children's intake of fruits and vegetables (FV) affect intake whether such effects are moderated by children's FV preferences and; we hypothesize that serving large fruit and vegetable portions will produce increases in children's intake of these foods, particularly for children who like fruit and vegetables. Experiment 3 will evaluate how food energy density affects children's response to large portions; we hypothesize that large portions will have the greatest influence on children's energy consumption when foods are energy dense. Experiment 4 will begin to address perceptual mechanisms by which large portions affect children's eating.

DETAILED DESCRIPTION:
The emerging epidemic of overweight among underscores the need to identify contributing environmental factors. Marketplace trends for excessive and growing portion sizes in and outside the home have reinforced concerns that large portions may directly contribute by promoting excessive intake. To date, however, systematic investigation of portion size effects on children's eating has been extremely limited. Two laboratory studies have reported that serving large portions of macaroni and cheese to young children promoted energy consumption at meals. Whether portion size effects would be seen with other foods of varying energy content and preference is unknown. Of particular public health interest is whether serving large portions may affect children's intake of sweetened beverages, fruits and vegetables, and energy dense foods. This study will address these questions using an experimental approach to test the effects of portion size on children's eating.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 6 years

Exclusion Criteria:

* severe food allergies
* chronic illnesses or medication use affecting food intake
* dislike of foods on the menu

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2005-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Intake of portion manipulated foods | In each experimental condition; 4 times in each 2 x 2 factorial experiment
Total energy consumed | In each experimental condition; 4 times in each 2 x 2 factorial experiment

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer O Fisher, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Center for Obesity Research, Temple University, Philadelphia, Pennsylvania
  - USDA\ARS Children's Nutrition Research Center, Houston, Texas